CLINICAL TRIAL: NCT04375930
Title: The Effect of Standard-Based Care on Peristomal Skin Complications and Quality of Life in Ostomy Creation Patients With Colorectal Cancer
Brief Title: Peristomal Skin Complications and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Cahide AYİK, Research assistant, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3491-GOA
Record Dates: First submitted 2020-01-27; First posted 2020-05-06 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer; Quality of Life; Stoma Ileostomy; Stoma Colostomy; Complication
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This two-group, single-blind, quasi-experimental study enrolled 68 patients with ostomy recruited to a university affiliated hospital.
Who Masked: Participant
Masking Description: The patients with an ostomy were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The patient will be trained with STANDARD STOMA CARE AND COMPLICATION DIAGNOSTIC ALGORITHM EDUCATION. The patient will be follow up at 2nd, 6th and 12th weeks.
  Interventions: Other: STANDARD STOMA CARE AND COMPLICATION DIAGNOSTIC ALGORITHM EDUCATION
- control (Active Comparator): The patient will be trained only skills and discharge education. The patient will be follow up at 2nd, 6th and 12th weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: STANDARD STOMA CARE AND COMPLICATION DIAGNOSTIC ALGORITHM EDUCATION — STANDARD STOMA CARE AND COMPLICATION DIAGNOSTIC ALGORITHM EDUCATION: It is consist of skills, discharge, compilation and algorithm education.
  Arms: Experimental
Other: Control — It consists of only skills and discharge education
  Arms: control

SUMMARY:
This study is a single blind semi-experimental study.

Aim: To investigate the effect of standardized care on peristomal skin complications and quality of life in colorectal cancer patients undergoing ostomy surgery.

H1: Standard stoma care which is established evidence-based guides and complication algorithm, reduces peristomal skin complications in patients with colorectal cancer and an ostomy.

H2: Standard stoma care which is established evidence-based guides and complication algorithm, increases the quality of life in patients with colorectal cancer and an ostomy.

DETAILED DESCRIPTION:
In order to ensure blindness in the study design, patients were not informed about which group they belonged to.

Patient with ostomy in the study group were trained in accordance with the Standard Stoma Care.

Patient with ostomy in the control group only skill and discharge training has been provided in accordance with the hospital procedure.

All patients were followed up at 2, 6, and 12 weeks. Peristomal complications were evaluated by the researcher with the Peristomal Skin Tool at the 2nd, 6th and 12th weeks. The patients were asked to fill the Stoma Quality of Life Scale in the 2nd, 6th and 12th weeks.

ELIGIBILITY:
Inclusion Criteria:

* undergoing colorectal surgery,
* permanent or temporary ileostomy or colostomy
* end or loop ileostomy or colostomy

Exclusion Criteria:

* individuals who have previously had stoma surgery,
* having two or more stoma,
* individuals with crohn's disease
* individuals who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of Peristomal skin complication change | 0, 2nd, 6th and 12th weeks
  It has been assessed with Ostomy Skin Tool. The total score can be the lowest 0 and the highest 15.
means of quality of life change | 2nd, 6th and 12th weeks
  It has been assessed with stoma Quality of Life Scale. The Scale range: 0-100. Higher scores for each item indicate that the quality of life increased.

CONTACTS AND LOCATIONS:
Overall Officials: Cahide Ayik, Principal Investigator — Dokuz Eylul University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)